CLINICAL TRIAL: NCT04371549
Title: Skin Closures at Cesarean Delivery, Glue vs Subcuticular Sutures: A Randomized Clinical Trial
Brief Title: Skin Closures at Cesarean Delivery, Glue vs Subcuticular Sutures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Elmaraghy, Lecturer of obstetrics and gynecology - faculty of medicine - Ainshams university, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Cesarean Wound; Dehiscence
MeSH Terms: interventions — Adhesives; octyl 2-cyanoacrylate; glycolide E-caprolactone copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glue (Active Comparator): Skin closure after cesarean section using glue
  Interventions: Procedure: Glue (Dermabond®; Ethicon, Somerville, NJ).
- Monocryl (Active Comparator): Skin closure after cesarean section using running subcuticular sutures using synthetic monofilament
  Interventions: Procedure: Monocryl

INTERVENTIONS:
Procedure: Glue (Dermabond®; Ethicon, Somerville, NJ). — Arm 1: Skin after cesarean section will be closed by glue
  Arms: Glue
Procedure: Monocryl — Arm 2: Skin after cesarean section will be closed by running subcuticular sutures using synthetic absorbable monofilament
  Arms: Monocryl

SUMMARY:
The optimal choice of skin closure at cesarean delivery has not yet been determined. This study will compare wound complications and scar healing following cesarean delivery between 2 methods of skin closure: glue (Dermabond®; Ethicon, Somerville, NJ) and monofilament (Monocryl®; Ethicon) epidermal sutures.

DETAILED DESCRIPTION:
Cesarean delivery (CD) rates have increased during the last few decades and it has become the most common surgery during women's reproductive years . However, despite its prevalence, data regarding many aspects of the preferred surgical technique are sparse. Skin closure is an integral step of CD. It influences postoperative pain, wound healing, cosmetic outcome, and surgeon and patient satisfaction There is currently no definite evidence regarding the best method for skin closure after cesarean delivery. Staples have been suggested as inferior to other techniques . Given the conflicting data available, obstetricians are forced to base their decisions on personal preference. Dermabond® glue (Ethicon Inc, Somerville, NJ) is a liquid monomer that forms a strong tissue bond with a protective barrier that adds strength and inhibits bacteria. An in vitro study found that glue inhibits both gram-positive (methicillin-resistant Staphylococcus aureus and Staphylococcus epidermidis) and gram-negative (Escherichia coli) bacteria . In addition, glue has the potential advantages of rapid application and repair time. It has been shown to achieve cosmetically similar results compared to staples within 12 months of the repair. Also, glue was shown to be well-accepted by patients .

To date, there have been no randomized clinical trials comparing skin closure with glue to sutures using the Patient and Observer Scar Assessment Scale (POSAS). The POSAS is a validated and reliable instrument that is practical for assessing scars . It is comprehensive and correlates well with patient ratings. The Observer Scar Assessment Scale rates 5 variables: vascularity, pigmentation, thickness, relief, and pliability. Each variable is ranked from 1-10, with 1 representing normal skin. Ratings are summed to obtain a total score ranging from 5-50. The Patient Scar Assessment Scale consists of 6 items: scar-related pain, itchiness, color, stiffness, thickness, and irregularity. Each item is ranked from 1-10, with 1 representing normal skin. Total score ranges from 6-60.

Previous studies regarding skin closure with glue were small, retrospective, and included mixed populations and varying surgical techniques. Therefore, clear, conclusive recommendations are lacking.

Dermabond® is a liquid monomeric (2-octyl cyanoacrylate) formulation that undergoes an exothermic reaction upon exposure to moisture, changing to polymers that form a strong tissue bond. The wound will not be dressed with an abdominal pad or adhesive tape according to manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* Maternal Age: 20-40 years old.
* BMI: 18.5 - 29.9 kg/m2.
* Gestational Age: term pregnancy (≥ 37 weeks) and viable fetus.
* Scheduled to undergo elective lower segment CD (category 4 CD).
* Hemoglobin level: ≥ 10 gm/dl.

Exclusion Criteria:

* Abnormal placental invasion (e.g., placenta previa).
* Emergency CD (category 1, 2 and 3 CD).
* Clinical signs of infection at the time of CD.
* Medical disorder (Diabetes, Hypertension, Cardiac, Hepatic or renal disorder).
* Uterine anomalies (e.g., septum, Mullerian anomalies or fibroids).
* Previous CD not using Pfannenstiel method (e.g., midline incision).
* Known hypersensitivity to any of the suture materials or glue used in the protocol, or any disorders requiring chronic corticosteroids or immune suppressants.
* History of surgical site infection after previous CD.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The Patient and Observer Scar Assessment Scale (POSASv2.0): | one week after cesarean section
  In the POSASv2.0 observers rate vascularity, pigmentation, pliability, thickness, relief and surface area. The directions for use of the different parameters of the Observer Scale POSASv2.0 are as follows (all parameters should be compared to normal skin at a comparable anatomical site whenever possible):The Patient Scale contains six questions applying to pain, itching, colour, pliability, thickness and relief.Each of the six items on both scales has a 10-point score, with 10 indicating the worst imaginable scar or sensation. The lowest score is '1' and corresponds to the situation of normal skin (normal pigmentation, no itching etc.), and goes up to the worst imaginable
The Patient and Observer Scar Assessment Scale (POSASv2.0): | one month after cesarean section
  In the POSASv2.0 observers rate vascularity, pigmentation, pliability, thickness, relief and surface area. The directions for use of the different parameters of the Observer scale POSASv2.0 are as follows ( all parameters should be compared to normal skin at a comparable anatomical site whenever possible): The Patient scale contains six questions applying to pain, itching, colour, pliability, thickness and relief. Each of the six items on both scales has a 10-point score, with 10 indicating the worst imaginable scar or sensation. The lowest score is 1 and correspons to the situation of normal skin( normal pigmentation, no itching etc.) and goes up to the worst imaginable

SECONDARY OUTCOMES:
Surgeons' satisfaction scale: | immediately after the procedure
  Surgeons' satisfaction scale with each closure method (glue vs sutures) is based on 3 questions asked immediately upon completion of surgery: (1) How comfortable were you with the technique? (not at all [1] to totally comfortable [5]); (2) Was the estimated total operating time longer using glue compared to skin closure with sutures? (not at all [1] to yes, a lot longer [5]); and (3) Were you satisfied with the final closure appearance? (not at all [1] to yes, very satisfied [5])
Duration of surgery | in minutes from closure of the subcutaneous fat layer to closure of the skin
  the duration of skin closure using glue or Monocryl will be measures in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud K Mohammed, M.B.B.Ch, Principal Investigator — AinShams university
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

REFERENCES:
- [Background] Altman R, Bosch B, Brune K, Patrignani P, Young C. Advances in NSAID development: evolution of diclofenac products using pharmaceutical technology. Drugs. 2015 May;75(8):859-77. doi: 10.1007/s40265-015-0392-z. PMID 25963327
- [Background] ACOG Practice Bulletin No. 199 Summary: Use of Prophylactic Antibiotics in Labor and Delivery. Obstet Gynecol. 2018 Sep;132(3):798-800. doi: 10.1097/AOG.0000000000002834. PMID 30134418
- [Background] Bhende S, Rothenburger S, Spangler DJ, Dito M. In vitro assessment of microbial barrier properties of Dermabond topical skin adhesive. Surg Infect (Larchmt). 2002 Fall;3(3):251-7. doi: 10.1089/109629602761624216. PMID 12542926
- [Background] Blanchette H. The rising cesarean delivery rate in America: what are the consequences? Obstet Gynecol. 2011 Sep;118(3):687-690. doi: 10.1097/AOG.0b013e318227b8d9. PMID 21860302
- [Background] Bruns TB, Worthington JM. Using tissue adhesive for wound repair: a practical guide to dermabond. Am Fam Physician. 2000 Mar 1;61(5):1383-8. PMID 10735344
- [Background] Clay FS, Walsh CA, Walsh SR. Staples vs subcuticular sutures for skin closure at cesarean delivery: a metaanalysis of randomized controlled trials. Am J Obstet Gynecol. 2011 May;204(5):378-83. doi: 10.1016/j.ajog.2010.11.018. Epub 2010 Dec 31. PMID 21195384
- [Background] Cromi A, Ghezzi F, Gottardi A, Cherubino M, Uccella S, Valdatta L. Cosmetic outcomes of various skin closure methods following cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2010 Jul;203(1):36.e1-8. doi: 10.1016/j.ajog.2010.02.001. Epub 2010 Apr 24. PMID 20417924
- [Background] Daykan Y, Sharon-Weiner M, Pasternak Y, Tzadikevitch-Geffen K, Markovitch O, Sukenik-Halevy R, Biron-Shental T. Skin closure at cesarean delivery, glue vs subcuticular sutures: a randomized controlled trial. Am J Obstet Gynecol. 2017 Apr;216(4):406.e1-406.e5. doi: 10.1016/j.ajog.2017.01.009. Epub 2017 Jan 30. PMID 28153666
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Siddiqui DS, Lacuna EM, Chen HY, Chauhan SP. Skin closure of pfannenstiel incision with dermabond, staples, or suture during cesarean delivery: experience of a single attending. Am J Perinatol. 2013 Mar;30(3):219-24. doi: 10.1055/s-0032-1323583. Epub 2012 Aug 8. PMID 22875661
- [Background] Singer AJ, Hollander JE, Quinn JV. Evaluation and management of traumatic lacerations. N Engl J Med. 1997 Oct 16;337(16):1142-8. doi: 10.1056/NEJM199710163371607. No abstract available. PMID 9329936
- [Background] Singer AJ, Quinn JV, Clark RE, Hollander JE; TraumaSeal Study Group. Closure of lacerations and incisions with octylcyanoacrylate: a multicenter randomized controlled trial. Surgery. 2002 Mar;131(3):270-6. doi: 10.1067/msy.2002.121377. PMID 11894031
- [Background] Truong PT, Lee JC, Soer B, Gaul CA, Olivotto IA. Reliability and validity testing of the Patient and Observer Scar Assessment Scale in evaluating linear scars after breast cancer surgery. Plast Reconstr Surg. 2007 Feb;119(2):487-94. doi: 10.1097/01.prs.0000252949.77525.bc. PMID 17230080
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683